CLINICAL TRIAL: NCT04136080
Title: The Effect of Increasing the Mean Arterial Pressure on the Microcirculation and the Prognosis of Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, Senior physician, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05-025
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic hypertension group (Other): septic patients with chronic hypertension
  Interventions: Other: vasopressors
- denying chronic hypertension group (Other): septic patients without chronic hypertension
  Interventions: Other: vasopressors

INTERVENTIONS:
Other: vasopressors — control the mean arterial pressure with vasopressors

SUMMARY:
Background： The mean arterial pressure（ MAP） is a key pressure index to improve tissue perfusion. At present, there are no surprising results of large-scale clinical studies on sublingual microcirculation. The changes of sublingual microcirculation were more severe in septic shock non-survivors than survivors. Purpose： This study is mean to increase the MAP in septic shock patients whether with chronic hypertension or not, so as to observe the change of the microcirculation and prognosis. Method： This is a single-center, randomized, prospective cohort study. Eligible patients will be allocated into chronic hypertension or denying chronic hypertension group. These patients will be treat with vasopressors to maintain MAP at 90±5 mmHg and 70±5 mmHg. Outcome： The 28-day all-cause mortality, the 90-day all-cause mortality, the 28-day without organ dysfunction days, the Changes of sublingual microcirculation, SOFA， APACHE-Ⅱ score Will be recorded.

ELIGIBILITY:
Adult patients (≥18 years) admitted to The Critical Medicine Departments Three of Fujian Provincial Hospital will be considered eligible，who are presence of infection or suspected infection，requiring mechanical ventilation. At the same time, without the vasopressors the MAP would be less than 65mmHg, and the blood lactic acid level is higher than 2mmol/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
the 28-day all-cause mortality and Changes of sublingual microcirculation | 28 day
  the 28-day all-cause mortality and Changes of sublingual microcirculation